CLINICAL TRIAL: NCT02987192
Title: Comparison of the Impact Between Minimally Invasive and Traditional Spinal Anesthesia for Cesarean Section in Maternal Anticoagulation Therapy:Randomized Controlled Trial
Brief Title: Minimally Invasive Lumbar Aneasthesia Used for Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, DAN HUANG, Dr., RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MICS2016033
Record Dates: First submitted 2016-11-16; First posted 2016-12-08 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Anticoagulation; Minimally Invasive; Spinal Anesthesia
Keywords: spinal anesthesia; anticoagulation; minimally invasive; Cesarean Section; Maternal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- traditional group (Experimental): Traditional group patients will receive cutting type 22 gauge needles
  Interventions: Device: cutting type 22 gauge needles
- minimally invasive group (Experimental): minimally invasive group patients will receive pen type 27 gauge needles
  Interventions: Device: pen type 27 gauge needles

INTERVENTIONS:
Device: pen type 27 gauge needles — minimally invasive group patients will receive pen type 27 gauge needles.
  Arms: minimally invasive group
Device: cutting type 22 gauge needles — traditional group patients will receive cutting type 22 gauge needles.
  Arms: traditional group

SUMMARY:
Spinal canal anesthesia is marked the most commonly used method of cesarean section. Traditional spinal anesthesia may cause post-dural puncture headache and low back pain.Plenty of parturients are undergoing anticoagulation therapy.They may be forced to accept general anesthesia in order to avoid epidural hematoma.Therefore, we propose minimally invasive spinal anesthesia.

DETAILED DESCRIPTION:
Traditional group patients will receive cutting type 22 gauge needles, while minimally invasive group patients will receive pen type 27 gauge needles.Patients will be blinded to the intervention allocations. Spinal anesthesia will be performed with a standardized technique. Lumbar puncture will be performed through an interspace (L3-4 or L2-3) with patients in a lateral decubitus position. After free flow of cerebrospinal fluid through the needle tip be verified, 2ml ropivacaine will be injected. We will record puncture situation, anesthesia plane and measure post-dural puncture headache, post-operative back pain and epidural hematoma.

ELIGIBILITY:
Inclusion Criteria:

1. puerpera accept anticoagulation therapy
2. American society of anesthesiologists(ASA) classification I to II level
3. Willing to participate in this study and signed an informed consent
4. pregnancy at least 37 weeks

Exclusion Criteria:

1. platelet count less than 50*100000000
2. International Normalized Ratio more than 1.5
3. site of puncture with infection
4. with intracranial hypertension
5. with lumbar spine or spinal cord disorders

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-07 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Visual analogue score of post-dural puncture headache | 1 to 7 days after operation

SECONDARY OUTCOMES:
Visual analogue score of low back pain | 1 to 7 days after operation

CONTACTS AND LOCATIONS:
Overall Officials: WEIFENG YU, MD, Study Chair — Anesthesiology Department Renji Hospital, Shanghai Jiao Tong University, School of Medicine
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Huang D, Zhu L, Chen J, Zhou J. Minimally invasive spinal anesthesia for cesarean section in maternal anticoagulation therapy: a randomized controlled trial. BMC Anesthesiol. 2019 Jan 12;19(1):11. doi: 10.1186/s12871-018-0679-1. PMID 30636632